CLINICAL TRIAL: NCT06419036
Title: The Use of Medical Devices to Monitor COPD Patients Study - An Observational Feasibility Study
Brief Title: The Use of Medical Devices to Monitor Chronic Obstructive Pulmonary Disease Patients Study BREATH-TRACHER 1
Acronym: BREATH-TRACHER
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Strathclyde (Other)
Collaborators: Pneumowave Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: UEC23/51
Record Dates: First submitted 2023-08-28; First posted 2024-05-17 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: COPD Exacerbation Acute
Keywords: medical device; remote monitoring technologies; respiratory signal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with COPD: The study population for this research consists of individuals diagnosed with COPD (Chronic Obstructive Pulmonary Disease) who have a history of exacerbation-induced hospitalization within the one-year period preceding recruitment.
  Interventions: Device: Pneumowave DC

INTERVENTIONS:
Device: Pneumowave DC — Pneumowave biosensor(s) will be used to collect data from chest +/- movement.

SUMMARY:
The proposed study will explore whether remote monitoring of a COPD patient can be undertaken using a wearable medical device.

DETAILED DESCRIPTION:
The proposed study will assess the sensitivity of a wearable device to measure the respiratory signals in COPD patients, who have previously experienced hospitalisation due to exacerbation of their COPD. Participation in the study involves wearing a small sensor. The monitoring device will also assess the effectiveness of medication prescribed before, during, and after the COPD exacerbation to see if it has a role in directing day-to-day therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any person aged 18 years or over.
* Current diagnosis of COPD.
* Be willing and able to comply with study procedures and be available for study visits. • Be able to use a 'smartphone or computer'.
* Be able to give written consent.
* Able to understand written and spoken English.

Exclusion Criteria:

* Inability to give written informed consent.
* Known respiratory disorders are other than COPD which, in the opinion of the investigator, is the main contributor to the patient's symptoms (e.g. asthma, lung cancer, sarcoidosis, and other interstitial lung diseases (ILDs), tuberculosis, lung fibrosis, cystic fibrosis, and non-COPD related bronchiectasis).
* Known history of significant systemic and other organ-related diseases, other than COPD, which in the opinion of the investigator, is likely to interfere with the study or impact on subject safety (e.g. severe rheumatoid arthritis and Lupus, kidney, liver, endocrine, psychological disorders).
* Known to be severely alpha-1-antitrypsin deficient (PI, SZ or ZZ).
* Based on their medical record if there is any social violence/substance misuse.
* Having undergone lung surgery (e.g. lung volume reduction, lobectomy) within the last 6 months.
* Have cancer or other terminal condition which, in the opinion of the investigator, has a mortality of 12 months or less. • Have, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse.
* Taking high-dose oral corticosteroid medication (equivalent to daily dose of ≥10 mg of prednisolone) for more than 3 consecutive months.
* Pregnancy
* Patients already involved in an ongoing research study.
* Participation in an interventional clinical study within 3 months of Visit 1 or participation in a study using an investigational medicinal product (IMP) either in the previous 3 months or in the interval from last using the IMP to 5 times its half-life.
* Patients with other significant lung disease, unable to consent, unable to use the technology (e.g. inability to use the data device, or complete the questionnaires), or at the clinician's discretion for other more significant medical/social reasons.
* Known allergy to surgical adhesive tape.
* On long-term oxygen therapy.
* Acute exacerbation of COPD within 6 weeks prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this research consists of individuals diagnosed with COPD (Chronic Obstructive Pulmonary Disease) who have a history of exacerbation-induced hospitalization within the one-year period preceding recruitment. The target number of participants in this study is 30.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical changes before COPD exacerbations | 18 months
  Participants' breath rates will be measured through chest movement in their daily lives, and clinical changes in their breath rates will be examined.

SECONDARY OUTCOMES:
Device usage | 18 months
  • To assess the usability and comfort of the wearable technology, assessed by qualitative interviews and field notes during fortnightly follow-up appointments from the perspective of the volunteer

CONTACTS AND LOCATIONS:
Locations (1):
- Oakview Medical Practice in Alexandria, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data collected during the study will be immediately anonymized and will not be shared with third parties.

REFERENCES:
- [Background] Hawthorne G, Richardson M, Greening NJ, Esliger D, Briggs-Price S, Chaplin EJ, Clinch L, Steiner MC, Singh SJ, Orme MW. A proof of concept for continuous, non-invasive, free-living vital signs monitoring to predict readmission following an acute exacerbation of COPD: a prospective cohort study. Respir Res. 2022 Apr 26;23(1):102. doi: 10.1186/s12931-022-02018-5. PMID 35473718
- [Background] Seemungal TA, Hurst JR, Wedzicha JA. Exacerbation rate, health status and mortality in COPD--a review of potential interventions. Int J Chron Obstruct Pulmon Dis. 2009;4:203-23. doi: 10.2147/copd.s3385. Epub 2009 Jun 11. PMID 19554195
- [Background] Donaldson GC, Law M, Kowlessar B, Singh R, Brill SE, Allinson JP, Wedzicha JA. Impact of Prolonged Exacerbation Recovery in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2015 Oct 15;192(8):943-50. doi: 10.1164/rccm.201412-2269OC. PMID 26151174